CLINICAL TRIAL: NCT03077646
Title: Pediatric Inpatient Firearm Safety Study
Acronym: IF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Collaborators: Everytown for Gun Safety (Other Government); Consano Clinical Research, LLC (Other)
Responsible Party: Principal Investigator, Alyssa Silver, Assistant Professor of Pediatrics, Attending Physician Pediatric Hospital Medicine, Montefiore Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2016-6918
Record Dates: First submitted 2017-01-31; First posted 2017-03-13 (Actual); Results first posted 2021-02-23 (Actual); Last update posted 2021-02-23 (Actual); Status verified 2021-02

CONDITIONS: Firearm Safety
Keywords: firearm; gun; safety; pediatric; inpatient

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Be SMART alone (Experimental): Parents/guardians in this study group will watch a 5.5 minute Be SMART video and receive the handouts reviewing the information.
  Interventions: Behavioral: Be SMART
- Be SMART + MD review (Experimental): Parents/guardians in this study group will watch a 5.5 minute Be SMART video and receive the handouts reviewing the information and will also have an MD review the information (via a checklist to standardize the MD review).
  Interventions: Behavioral: Be SMART + MD review
- Control: TSE materials (Active Comparator): Parents/guardians in this study group will watch a video "Kids and Smoke Don't Mix" and receive handouts reviewing information on tobacco smoke exposure (TSE).
  Interventions: Behavioral: Control: TSE

INTERVENTIONS:
Behavioral: Be SMART — An educational campaign that is non-political reviewing gun safety measures for preventing firearm injuries in children. There is both a video and written materials reviewing the information. The acronym SMART stands for: Secure all guns in your home, Model responsible behavior, Ask about unsecured guns in other homes, Recognize the risks of teen suicide, Tell your peers to be SMART
  Arms: Be SMART alone
Behavioral: Control: TSE — A video called "Kids and Smoke Don't Mix" and handouts on tobacco smoke exposure (TSE) developed by the New York state quit-line.
  Arms: Control: TSE materials
Behavioral: Be SMART + MD review — An educational campaign that is non-political reviewing gun safety measures for preventing firearm injuries in children. There is both a video and written materials reviewing the information. The acronym SMART stands for: Secure all guns in your home, Model responsible behavior, Ask about unsecured guns in other homes, Recognize the risks of teen suicide, Tell your peers to be SMART.
  After being presented to parents/guardians via video and handouts, this information will be reviewed in person with a Physician.
  Arms: Be SMART + MD review

SUMMARY:
There is currently no available data regarding using the inpatient setting as an opportunity to talk to parents/guardians about firearm safety. The investigators will be doing a pre-/post-intervention study to investigate the effect of an intervention (a 5.5 minute Be SMART video and written materials developed by the organization Everytown for Gun Safety), on parental/legal guardian knowledge, attitudes and practices regarding firearm safety. While the American Academy of Pediatrics recommends the safest home for children is one without guns, the reality is that there are families with guns in the home. This non-political video focuses on ways to keep children safe from firearms.

The investigators will also investigate any additional effect of physician-delivered counseling on parental/guardian knowledge, attitudes and practices regarding gun safety as compared to receiving the information solely via video and written materials.

Participants will be randomized to 1 of 3 groups (intervention, intervention + MD discussion and control group). Outcomes will be assessed immediately post intervention and in a 30-day follow up phone call.

DETAILED DESCRIPTION:
Eligibility:

All parents/guardians of inpatients admitted to the Children's Hospital at Montefiore.

Exclusion:

Parents/guardians whose children are in acute distress or in the Pediatric Intensive Care Unit.

Outcomes:

The primary outcome is the change in parent/legal guardian's behavior over the past 30 days with respect to how often they asked whether or not there are guns in the home when their child/children goes to play in another's person's home, as indicated by a Likert scale assignment of an ordinal value (1-5, 1= never, 2=rarely, 3=sometimes, 4=most of the time, 5=always).

Secondary outcomes will include:

* Change in the primary outcome (intention to ask noted above) between the intervention groups (Be SMARTalone vs. Be SMART + MD)
* Demographic factors associated with primary outcome
* Description of general knowledge on firearm safety of parents/legal guardians of patients in our community
* Description of attitudes about firearm safety of parents/legal guardians of patients in our community
* Description of general practices regarding firearm safety of parents/legal guardians of patients in our community
* Description of parents attitudes regarding physicians discussing firearm safety with them

ELIGIBILITY:
Inclusion Criteria:

-

Exclusion Criteria:

* parents/guardians whose child is hospitalized in the Pediatric Intensive Care Unit
* parents/guardians whose child is in acute distress
* parents/guardians who have previously been in the study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 225 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2019-08-09 (Actual); Study Completion 2019-08-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alyssa H Silver, MD, Principal Investigator — Children's Hospital at Montefiore-Department of Pediatrics, Division of Hospital Medicine
Locations (1):
- Children's Hospital at Montefiore, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share individual participant data with other researchers. The data will only be available to study personnel approved on this study.

REFERENCES:
- [Derived] Silver AH, Curley M, Azzarone G, Dodson N, O'Connor K. A Parent Survey Assessing Association of Exposure to Gun Violence, Beliefs, and Physician Counseling. Hosp Pediatr. 2022 Mar 1;12(3):e95-e111. doi: 10.1542/hpeds.2021-006050. PMID 35112128
- [Derived] Silver AH, Azzarone G, Dodson N, Curley M, Eisenberg R, Kim M, O'Connor K. A Randomized Controlled Trial for Parents of Hospitalized Children: Keeping Kids Safe From Guns. Hosp Pediatr. 2021 Jul;11(7):691-702. doi: 10.1542/hpeds.2020-001214. Epub 2021 Jun 23. PMID 34162699

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study examine knowledge, attitudes, and practices of parents/legal guardians regarding firearm safety and tobacco smoke exposure. Children were not enrolled.
Pre-assignment Details: The parent/guardian only was enrolled (child was not), therefore it is not a dyad.
Groups:
- Be SMART + MD Review: Parents/guardians in this study group will watch a 5.5 minute Be SMART video and receive the handouts reviewing the information and will also have an MD review the information (via a checklist to standardize the MD review).
  Be SMART + MD review: An educational campaign that is non-political reviewing gun safety measures for preventing firearm injuries in children. There is both a video and written materials reviewing the information. The acronym SMART stands for: Secure all guns in your home, Model responsible behavior, Ask about unsecured guns in other homes, Recognize the risks of teen suicide, Tell your peers to be SMART.
  After being presented to parents/guardians via video and handouts, this information will be reviewed in person with a Physician.
Period: Overall Study
Arm/Group | Be SMART Alone | Be SMART + MD Review | Control: TSE Materials
Started | 76 | 75 | 74
Completed | 47 (Of these 47, there were 25 paired samples for primary outcome) | 45 (Of these 45, there were 27 paired samples for primary outcome) | 43 (Of these 43, there were 20 paired samples for primary outcome)
Not Completed | 29 | 30 | 31
Not completed — Lost to Follow-up | 29 | 30 | 31

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Be SMART Alone | Be SMART + MD Review | Control: TSE Materials | Total
Number analyzed (Participants) | 76 | 75 | 74 | 225
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 34.0 [27.5 to 41.0] | 35.0 [30.0 to 40.0] | 32.0 [27.0 to 38.0] | 33.0 [28.0 to 40.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 65 | 66 | 65 | 196
  Male | 11 | 9 | 9 | 29
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Child Race/ethnicity: Hispanic | 39 | 42 | 45 | 126
  Child Race/ethnicity: Non-Hispanic Black | 29 | 19 | 20 | 68
  Child Race/ethnicity: Non-Hispanic White | 2 | 3 | 5 | 10
  Child Race/ethnicity: Other | 6 | 11 | 4 | 21
Child age (years), median (IQR) [Median (Inter-Quartile Range); unit: years] | 4.5 [1.1 to 12.0] | 6.0 [1.0 to 12.0] | 4.0 [0.9 to 10.0] | 5.0 [1.0 to 11.0]
Child gender [Count of Participants; unit: Participants]
  Male | 33 | 48 | 34 | 115
  Female | 43 | 26 | 40 | 109
  Missing | 0 | 1 | 0 | 1
Parental education [Count of Participants; unit: Participants]
  Elementary school | 1 | 2 | 2 | 5
  Some High school | 8 | 6 | 8 | 22
  High School | 34 | 32 | 36 | 102
  College | 28 | 27 | 23 | 78
  Graduate school | 5 | 8 | 5 | 18
Language [Count of Participants; unit: Participants]
  English | 73 | 67 | 71 | 211
  Spanish | 3 | 6 | 3 | 12
  Mixed English & Spanish | 0 | 2 | 0 | 2
Insurance [Count of Participants; unit: Participants]
  Private | 26 | 22 | 15 | 63
  Medicaid | 46 | 49 | 55 | 150
  None | 2 | 0 | 2 | 4
  Other | 2 | 1 | 0 | 3
  Missing | 0 | 3 | 2 | 5
Seen a person with a gun? [Count of Participants; unit: Participants] | 23 | 24 | 18 | 65
Heard gunshots in your neighborhood [Count of Participants; unit: Participants] | 51 | 42 | 42 | 135
Raised in a home with a gun? [Count of Participants; unit: Participants] | 4 | 8 | 2 | 14
Been threatened with a gun? [Count of Participants; unit: Participants] | 6 | 8 | 7 | 21
Been shot with a gun? [Count of Participants; unit: Participants] | 1 | 1 | 1 | 3
Have a friend/relative shot with a gun? [Count of Participants; unit: Participants] | 39 | 27 | 28 | 94
Friend or relative has a gun? [Count of Participants; unit: Participants] | 21 | 20 | 18 | 59
Child has seen a gun? [Count of Participants; unit: Participants] | 5 | 6 | 4 | 15
Child has touched a gun? [Count of Participants; unit: Participants] | 2 | 3 | 2 | 7
Discussed with child what to do if they find a gun? [Count of Participants; unit: Participants] | 19 | 17 | 17 | 53
Discussed with other children what do do if they find a gun? [Count of Participants; unit: Participants] | 21 | 23 | 22 | 66
Guns have been brought into your home by guests [Count of Participants; unit: Participants] | 7 | 7 | 5 | 19
Have a gun in your home [Count of Participants; unit: Participants] | 4 | 2 | 2 | 8
Worry your child would play with a gun if they find one [Count of Participants; unit: Participants] | 45 | 41 | 42 | 128
Child's doctor has ever talked about gun safety [Count of Participants; unit: Participants] | 5 | 9 | 4 | 18
For those who don't have a gun, you would feel safer if you had a gun [Count of Participants; unit: Participants] | 7 | 7 | 4 | 18
It is important to ask about guns in others' homes when your child goes there [Mean (Standard Deviation); unit: Likert score scale of agreement (1-5)] | 4.4 (1) | 4.3 (1) | 4.4 (1) | 4.3 (0.7)

OUTCOME MEASURES:

1. Primary Outcome: Change in Likert Scale of Frequency of Asking About Guns in the Home When Their Child Goes to Another Person's Home, Pre-intervention and 1 Month Post-intervention
Description: The primary outcome is within each group the change in how often the parent/guardian asked whether there are guns in the home when the child went to another person's home in the last 30 days Likert Scale 1=never, 2=rarely, 3=sometimes, 4=most of the time, 5=always
Time Frame: Baseline and last 30 days
Population: Limited sample for analysis to paired samples within each group (samples where we have responses from the same study subject pre and post)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Be SMART Alone | Be SMART + MD Review | Control: TSE Materials
Number analyzed (Participants) | 25 | 27 | 20
score on a scale | 0.8 (1.7) | 0.6 (1.3) | 0.9 (1.4)

2. Secondary Outcome: Doctors Who Take Care of Kids Should Talk to Parents About Safe Gun Storage at 1 Month Post-intervention
Description: Likert Scale Score of degree of agreement with the statement
  1=strongly disagree, 2=disagree, 3=not sure, 4=agree, 5=strongly agree
Time Frame: 1 month after intervention
Population: Some parents unable to reach by phone at 1 month
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Be SMART Alone | Be SMART + MD Review | Control: TSE Materials
Number analyzed (Participants) | 47 | 44 | 43
score on a scale | 4.2 (0.9) | 4.3 (0.8) | 4.3 (0.8)

ADVERSE EVENTS:
Time Frame: One month
Description: No events reported for this educational intervemtion
Arm/Group | Be SMART Alone | Be SMART + MD Review | Control: TSE Materials
All-Cause Mortality (participants affected / at risk) | 0/76 | 0/75 | 0/74
Serious Adverse Events (participants affected / at risk) | 0/76 | 0/75 | 0/74
Other Adverse Events (participants affected / at risk) | 0/76 | 0/75 | 0/74

LIMITATIONS AND CAVEATS:
Single center with particular "gun culture" may not be generalizable to other regions of the country.

Limited paired sample follow-up, therefore may be underpowered.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-01-20): https://cdn.clinicaltrials.gov/large-docs/46/NCT03077646/Prot_SAP_000.pdf